CLINICAL TRIAL: NCT06838234
Title: Validity and Reliability of Arabic Version of the Quality of Life Questionnaire in Patients With Chronic Wound
Brief Title: Arabic Version QOL Questionnaire Chronic Wound
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Harown Boshra Eskandar, Physiotherapist at 23rd of July hospital,M.SC physiotherapy, Cairo university, Cairo University
Other Study IDs: P.T.REC/012/024127
Record Dates: First submitted 2025-02-09; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chronic Wound
Keywords: Validity and reliability. .; Arabic version QOL questionnaire; chronic wound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 group suffering from chronic wound: Patients who have chronic wound will answer the items of the questionnaire
  Interventions: Other: Arabic version QOL questionnaire

INTERVENTIONS:
Other: Arabic version QOL questionnaire — Arabic version QOL questionnaire The Wound-QoL is a wound-specific questionnaire containing 17 items from which one can derive three subscales and . The items 1-5, 6-10, and 11-16 belong to the subscale body, psyche, and everyday life, respectively

SUMMARY:
The aim of this study is to Help clinician modification of treatment through assess the validity and reliability of Arabic version of 17 items QOL questionnaire in patients with chronic wound. It translated to many languages but not present in form of arabic version.

DETAILED DESCRIPTION:
The study will be cross sectional.participants: 100 patients according to sample size calculations suffering from chronic wound with age between 40-60 years. Using the minimum acceptable ICC of 0.75, expected ICC of 0.85, significance level 0.05, statistical power 80% and number of repetitions 2, the required sample size is about 100 subjects.The patients who met the inclusion criteria will be recruited. The purpose, significance, and procedures of the study will be explained to them, and written informed consent Will be obtained before enrollment.The researcher will measure the wounds and collect disease-related data during dressing changes. The participants will then be asked to fill out the questionnaires by themselves or with the help of the researcher.Each item is scored on a 5-point Likert scale from 0 (not at all) to 4 (very much). On obtaining at least 75% response, the researcher calculated a second-order global score as well as scores for every dimension as the mean of the respective responses. Higher scores indicated greater impairment of the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffering from chronic wound at least 1 month prior to study enrollment,
* Patients aged between 40-60 years .Provision of written informed consent. .All participants will be able to read and write in Arabic language. .All participants can understand items of the questionnaire.

Exclusion Criteria:

* Patients who had mental illnesses
* Patients who were unable to fill in the questionnaire independently or answered the questions orally .Patient with communication, vision, hearing disorders. .Patient who doesn't fill the questionnaire till the end.
* Patient who were isolated due to infection

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study includes 100 patients of both sexes with chronic wound with ages between 40-60 years. Recruited from outpatient clinic of Faculty of Physical Therapy Cairo University and El matarya hospital Patients with chronic wound at least one month ( Venus and arterial ulcer , diabetic foot, burn , Post operative wound healing defect)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Body subscale | outcome measure will be applied after one month of wound injury
  Body subscale include items (1-5). (My wound hurt, my wound had a bad smell , there was a distributing discharge from wound, the wound has affected my sleep , the treatment of the wound has been burden to me) score range from 0 to 4 , score 0 indicate better and score 4 indicate worser
Psyche subscale | outcome measure will be applied after one month of wound injury
  Psyche subscale include items (6_10), score range from 0 to 4 , score 0 indicate better and score 4 indicate worser ( The wound has made me unhappy, I have felt frustrated because the wound is taking so long to heal, I have worried about my wound,I have afraid of the wound getting worse or of new wounds appearing,I have afraid of knocking the wound
Day life subscale | outcome measure will be applied after one month of wound injury
  Day life subscale include items (11-16)I have been a trouble moving about because of the wound, climbing stairs has been difficult because of the wound, I have had a trouble with day to day activities , The wound has limited my leisure activities , The wound has forced me to limit activities with others, I have felt dependant on help from other. score range from 0 to 4 , score 0 indicate better and score 4 indicate worser

CONTACTS AND LOCATIONS:
Overall Officials: Karim I Abo Khalil safaan, Principal Investigator — Assistant Professor at surgery and burn Department , Faculty of Physical Therapy Cairo University
Locations (1):
- Cairo University, Cairo, Egypt